CLINICAL TRIAL: NCT03080818
Title: Evaluation of a Probiotic on Psychological and Cognitive Effects in Middle and Older Adults
Brief Title: Probiotic on Psychological and Cognitive Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: iHealth (Other)
Responsible Party: Principal Investigator, John Gunstad, Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Kent State University
Record Dates: First submitted 2017-03-05; First posted 2017-03-15 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Aging
Keywords: Probiotic, Cognitive Function, Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants in this arm will receive probiotic supplementation for 12 weeks (Lactobacillus Rhamnosus GG)
  Interventions: Dietary Supplement: Probiotic - Lactobacillus Rhamnosus GG
- Control (Placebo Comparator): Participants in this arm will receive placebo that look similar to probiotics
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic - Lactobacillus Rhamnosus GG — 2 capsules per day for 90 days
  Arms: Probiotic
Other: Placebo — 2 placebo capsules per day for 90 days
  Arms: Control

SUMMARY:
This study will determine whether supplementation of probiotic Lactobacillus Rhamnosus GG improves psychological status in middle age and older adults through a 12-week, randomized, double-blind, placebo-controlled clinical trial. Secondary analyses will be conducted to examine the possible benefits of probiotic supplementation on cognitive function and markers of physical health.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-75 years
* Able to speak and read English

Exclusion Criteria:

* History of neurological, developmental, or severe psychiatric disorder (e.g. dementia, stroke, schizophrenia);
* Antibiotic use in the past 30 days;
* History of significant stomach or GI surgery (e.g. gastric bypass, cholecystectomy);
* History of alcohol or illicit drug dependence;
* History of severe heart, kidney, or liver problems (e.g. heart failure, liver failure);
* Regular use of an acid-blocking medication in the past 30 days (i.e. proton pump inhibitor, H2 blocker);
* Likely immunosuppression (e.g. chemotherapy treatment);
* Regular use of other pre- or probiotic supplements in the past 30 days;
* Severe gastrointestinal conditions including celiac disease, Crohn's disease, or diverticulitis.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in score on Center for Epidemiologic Studies Depression - R (CES-D-R) | Baseline and 12 week follow up
  Depressive symptoms
Change in score on State-Trait Anxiety Inventory | Baseline and 12 week follow up
  Anxiety symptoms
Change in score on Perceived Stress Scale | Baseline and 12 week follow up
  Subjective stress
Change in score on Positive and Negative Affect Schedule | Baseline and 12 week follow up
  Fluctuations in affect
Change in score on Profile of Mood States | Baseline and 12 week follow up
  Fluctuations in affect - acute
Change in score on Warwick-Edinburgh Mental Well-Being Scale | Baseline and 12 week follow up
  Subjective wellbeing
Change in score on OECD Life Satisfaction scale (short) | Baseline and 12 week follow up
  Subjective wellbeing - general
Change in score on Response to Stressful Events Scale | Baseline and 12 week follow up
  Emotion regulation
Change in score on Connor-Davidson Resilience Scale | Baseline and 12 week follow up
  Emotional resilience

SECONDARY OUTCOMES:
Change in Picture Sequence Memory Test and Auditory Verbal Learning Test scores | Baseline and 12 week follow up
  Memory
Change in Dimension Card Sort Test, Flanker Inhibitory Control, and List Sorting Working Memory Test scores | Baseline and 12 week follow up
  Executive function/Attention
Change in Pattern Comparison Processing Speed Test scores | Baseline and 12 week follow up
  Processing Speed
Change in SF-36 scores | Baseline and 12 week follow up
  Quality of Life
Change in Pittsburgh Sleep Quality Index scores | Baseline and 12 week follow up
  Sleep patterns
Change in Gastrointestinal Symptom Rating Scale scores | Baseline and 12 week follow up
  Subjective gastrointestinal symptoms
Change in HbA1c and fasting glucose values | Baseline and 12 week follow up
  Laboratory measures of glycemic control
Change in C-reactive protein, Interleukin-6, and TNF-alpha values | Baseline and 12 week follow up
  Laboratory measures of inflammation
Change in Total Cholesterol, HDL, LDL, and VLDL values | Baseline and 12 week follow up
  Laboratory meausres of lipid levels
Change in waking cortisol levels | Baseline and 12 week follow up
  Laboratory measure of cortisol
Change in composition of the gut microbiome | Baseline and 12 week follow up
  Laboratory measure of gut microbiome
Change in oral microbiome composition | Baseline and 12 week follow up
  Laboratory measure of oral microbiome

CONTACTS AND LOCATIONS:
Overall Officials: John Gunstad, Ph.D., Principal Investigator — Kent State University
Locations (1):
- Kent State Uniersity, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aljumaah MR, Bhatia U, Roach J, Gunstad J, Azcarate Peril MA. The gut microbiome, mild cognitive impairment, and probiotics: A randomized clinical trial in middle-aged and older adults. Clin Nutr. 2022 Nov;41(11):2565-2576. doi: 10.1016/j.clnu.2022.09.012. Epub 2022 Sep 28. PMID 36228569
- [Derived] Sanborn V, Aljumaah M, Azcarate-Peril MA, Gunstad J. Examining the cognitive benefits of probiotic supplementation in physically active older adults: A randomized clinical trial. Appl Physiol Nutr Metab. 2022 Aug 1;47(8):871-882. doi: 10.1139/apnm-2021-0557. Epub 2022 May 26. PMID 35617704